CLINICAL TRIAL: NCT00183157
Title: RAP: Reaching Adolescents for Prevention - A Randomized Trial of a Brief Negotiated Interview and Active Referral to Reduce Alcohol Related Morbidity Among Youth and Young Adults in the Pediatric Emergency Department
Brief Title: Project RAP: Reaching Adolescents for Prevention
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Edward Bernstein, MD/Judith Bernstein, RNC, PhD, Boston University School of Public Health - Youth Alcohol Prevention Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIAAABER13759; NIH 5P60 AA13759
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Alcohol Related Morbidity; Alcohol Dependence
Keywords: High risk drinking; Alcohol dependence; Alcohol related injury
MeSH Terms: conditions — Alcoholism | interventions — Restraint, Physical

ARMS (3):
- 1 (Active Comparator): Patients will receive an assessment, a brief motivational interview performed by a trained peer counselor, direct referrals to community-based resources for adolescents, and a 10-day follow-up phone call.
  Interventions: Behavioral: Brief Motivational Intervention
- 2 (Active Comparator): Patients will receive an assessment and a list of community resources
  Interventions: Behavioral: Assessment and list of resources
- 3 (Active Comparator): Patients will receive only the list of resources.
  Interventions: Behavioral: Referral to Community Resources

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — One-third of the enrollees will receive an assessment, a brief motivational interview performed by a trained peer counselor, direct referrals to community-based resources for adolescents, and a 10-day follow-up phone call. All participants will be followed over time and re-screened to measure the impact of the initial brief intervention on their drinking and drug-taking. The key hypothesis is that individuals who receive the brief motivational interview in the emergency department setting will have lower rates of alcohol and illicit drug use and fewer health consequences over time.
  Arms: 1
Behavioral: Assessment and list of resources — One-third will receive only the assessment and a list of community resources. All participants will be followed over time and re-screened to measure the impact of the initial brief intervention on their drinking and drug-taking. The key hypothesis is that individuals who receive the brief motivational interview in the emergency department setting will have lower rates of alcohol and illicit drug use and fewer health consequences over time.
  Arms: 2
Behavioral: Referral to Community Resources — All patients aged 14 to 21 get a brief alcohol and drug screen, and those whose scores indicate they drink or use marijuana are invited to participate in the study. One-third of the enrollees will receive only a list of resources. All participants will be followed over time and re-screened to measure the impact of the initial brief intervention on their drinking and drug-taking. The key hypothesis is that individuals who receive the brief motivational interview in the emergency department setting will have lower rates of alcohol and illicit drug use and fewer health consequences over time.
  Arms: 3

SUMMARY:
The purpose of the study is to determine if a brief motivational interview in the context of an emergency health care visit will reduce high-risk drinking and drug-taking and associated health consequences among adolescents ages 14-21 years old.

DETAILED DESCRIPTION:
Many studies have shown that a brief motivational interview in the context of a routine or emergency health care visit may assist adults to reduce high-risk drinking and drug-taking. Center researchers are conducting a 1,400-person, randomized clinical trial involving teen patients at the Boston Medical Center Pediatric Emergency Department in order to determine if a similar approach will be effective with youth. All patients aged 14 to 21 get a brief alcohol and drug screen, and those whose scores indicate they drink or use marijuana are invited to participate in the study. One-third of the enrollees will receive an assessment, a brief motivational interview performed by a trained peer counselor, direct referrals to community-based resources for adolescents, and a 10-day follow-up phone call. One-third will receive only the assessment and a list of community resources; and the final third will receive only the list of resources. All participants will be followed over time and re-screened to measure the impact of the initial brief intervention on their drinking and drug-taking. The key hypothesis is that individuals who receive the brief motivational interview in the emergency department setting will have lower rates of alcohol and illicit drug use and fewer health consequences over time.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric emergency department patients
* Aged 14-21
* An Alcohol Use Disorders Identification Test (AUDIT) score above selected cut-point for age or with history of alcohol-related consequences

Exclusion Criteria:

* Not resident in area or able to provide contact information for 12 month follow-up
* Medically unstable
* Not oriented to person, time and place

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2004-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in drinking | 12 months

SECONDARY OUTCOMES:
Reduction in alcohol associated health consequences | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bernstein, MD, Principal Investigator — Boston University School of Public Health - Youth Alcohol Prevention Center; Judith Bernstein, RNC, PhD, Principal Investigator — Boston University School of Public Health - Youth Alcohol Prevention Center
Locations (2):
- United States (2):
  - Boston Medical Center Pediatric Emergency Department, Boston, Massachusetts
  - Boston University School of Public Health - Youth Alcohol Prevention Center, Boston, Massachusetts

REFERENCES:
- See also: Reaching Adolescents for Prevention (RAP), Boston University School of Public Health — http://sph.bu.edu/index.php?option=com_content&task=view&id=412&Itemid=515